CLINICAL TRIAL: NCT05027984
Title: An Interventional Strategy for Non-culprit Lesions With Major Vulnerability Criteria Identified by Optical Coherence Tomography in Patients With Acute Coronary Syndrome (the INTER-CLIMA Trial)
Brief Title: Interventional Strategy for Non-culprit Lesions With Major Vulnerability Criteria at OCT in Patients With ACS
Acronym: INTERCLIMA
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centro per la Lotta Contro l'Infarto - Fondazione Onlus (Other)
Collaborators: Abbott Vascular (Santa Clara, USA) (Unknown)
Responsible Party: Principal Investigator, Francesco Prati, President of Centro per la Lotta Contro l'Infarto - Fondazione Onlus, Centro per la Lotta Contro l'Infarto - Fondazione Onlus
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CLI-01-2020
Record Dates: First submitted 2021-07-10; First posted 2021-08-31 (Actual); Last update posted 2025-07-28 (Actual); Status verified 2025-07

CONDITIONS: Coronary Artery Disease; Coronary Disease; Ischemic Heart Disease
Keywords: Coronary artery disease; Optical coherence tomography; Vulnerable plaque
MeSH Terms: conditions — Coronary Artery Disease; Coronary Disease; Myocardial Ischemia | interventions — Tomography, Optical Coherence

STUDY DESIGN:
Intervention Model Description: Two groups: one group receiving functional assessment of intermediate coronary lesions and the other group undergoing OCT assessment.
Who Masked: Outcomes Assessor
Masking Description: All events included in the study endpoints will be adjudicated by a blinded Clinical Event Adjudication Committee.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Intermediate lesion OCT-based management (Experimental): At OCT analysis, lesion features prompting intervention instead of conservative approach will be the following:
  1. FCT <75 µm, plus at least 2 of 3 other OCT criteria of plaque vulnerability (i.e., MLA <3.5 mm2, lipid arc with circumferential extension >180°, and the presence of macrophages).
  2. The presence of intracoronary thrombus at a non-culprit site, irrespective of the presence of other vulnerability criteria, may prompt treatment with DES, at the operator's discretion.
  All lesions fulfilling these interventional criteria will be treated with an OCT guided DES implantation in order to achieve an optimal stent implantation.
  In presence of a MLA <2.0 mm2, best cut-off showing correlation with fractional-flow reserve positive functional (FFR) assessment, clinical decision whether to treat the lesion will be based on FFR assessment irrespective of the presence of other criteria of vulnerability. Alternatively authors will have the option to treat the lesion with a DES.
  Interventions: Device: Optical coherence tomography
- Intermediate lesion physiology-based management (Active Comparator): The iFR/FFR/RFR measurements will be obtained using a coronary-pressure guidewire. For FFR, hyperemia will be induced with the administration of intravenous adenosine, in accordance with the clinical practice at each participating center. Lesion features prompting intervention instead of conservative medical approach will be the following: iFR ≤0.89, or FFR ≤0.80.(32) All lesions fulfilling these interventional criteria will be treated with an FFR guided DES implantation. PCI will be performed with the aim of achieving a post-stenting FFR ≥0.90 (i.e. optimal FFR result). If post-stenting FFR was <0.90 a further post-dilation of the stent could be performed and if FFR remained at <0.90, a pullback of the wire to identify another possible pressure drop and/or a subsequent stent implantation at least 5 mm from the stent will be performed according to physician's preference.
  Interventions: Device: iFR/FFR/RFR

INTERVENTIONS:
Device: Optical coherence tomography — OCT images will be acquired by means of the FD C7 XR system or the OPTIS system (both St. Jude Medical, St. Paul, MN, USA) with a non-occlusive technique.(33) The acquired OCT coronary images will be analyzed on-line using a proprietary OCT console (St Jude Medical, Inc., USA). Definitions and cut-offs for OCT vulnerability parameters derived from available consensus documents and from main IVUS/OCT studies.
  Arms: Intermediate lesion OCT-based management
Device: iFR/FFR/RFR — The iFR and FFR measurements will be obtained using a coronary-pressure guidewire (Pressure Wire / Certus or Aeris for FFR assessment and PressureWire™ X Guidewire/QUANTIEM™ for the RFR assessment by Abbott Vascular, Abbott Park, Illinois, U.S.A; Comet by Boston Scientific, Marlborough, MA, USA), OptoWire by Opsens, Quebec, Canada, or Verrata by Philips, San Diego, CA, USA.).
  Arms: Intermediate lesion physiology-based management

SUMMARY:
The INTERCLIMA (Interventional Strategy for Non-culprit Lesions With Major Vulnerability Criteria Identified by Optical Coherence Tomography in Patients With Acute Coronary Syndrome) is a multi-center, prospective, randomized trial of optical coherence tomography (OCT)-based versus physiology-based (i.e. fractional flow reserve[FFR]/instantaneous Wave-Free Ratio[iFR]/resting full-cycle ratio[RFR]) treatment of intermediate (40-70% diameter stenosis), non-culprit coronary lesions in acute coronary syndrome (ACS) patients undergoing coronary angiography. About 1420 patients with ACS will be randomized into the study at approximately 40 sites worldwide.

DETAILED DESCRIPTION:
The optimal strategy in patients with intermediated stenosis (40-70% diameter stenosis) at coronary angiography is currently under debate. Pure angiographic stenosis evaluation is often inadequate and alternative assessments of coronary plaques entered the clinical practice, such as functional assessment (FFR/iFR/RFR) and intravascular imaging (OCT and intravascular ultrasound [IVUS]). Based on preliminary data, current American College of Cardiology (ACC) and American Heart Association (AHA) revascularization guidelines recommend the use of flow fractional reserve (FFR, class IIa of evidence) to assess angiographic intermediate coronary lesions in patients with stable ischemic heart disease and guide intervention. However, controversial data has recently emerged on the role of functional assessment of intermediate coronary lesions in both acute and chronic settings. On the other hand, in recent studies, the presence of coronary plaques with vulnerability criteria at OCT identified patients at high risk of cardiac mortality and target vessel MI. This study aims to assess the clinical effectiveness of an OCT-based strategy to guide revascularization in non-culprit intermediate coronary stenosis in patients with acute coronary syndrome (ACS), on the basis of the presence of morphological markers of plaque vulnerability. Patients with intermediate coronary lesions in non-culprit intervention-naïve major coronary segments (diameter ≥2.5 mm) and fulfilling all inclusion/exclusion criteria will be eligible. Enrolled patients will be randomized 1:1 to either OCT or FFR/RFR/iFR based treatment. In the OCT-guided arm, non-culprit intermediate lesions will be treated with PCI with implantation of a second-generation drug eluting stent (DES) when a FCT <75 µm plus at least 2 of 3 other OCT criteria of plaque vulnerability (i.e., MLA <3.5 mm2, lipid arc with circumferential extension >180°, and the presence of clusters of macrophages) and/or an MLA <2 mm2 are detected by OCT. In the absence of the above-mentioned 4 vulnerability criteria, interventional procedures will be performed at discretion of the operator if a luminal thrombus is detected by OCT. In the physiology-guided arm, non-culprit intermediate lesions will be treated with PCI with implantation of a second-generation DES when an iFR or RFR ≤0.89 or an FFR ≤0.80 are measured, otherwise interventional procedures will be deferred. The primary endpoint, a composite of cardiac death and target vessel spontaneous myocardial infarction, will be assessed after 2 and 5 years.

ELIGIBILITY:
Inclusion Criteria:

* Age of at least 18 years.
* Diagnosis of acute coronary syndrome.
* Single or multiple intermediate lesions in intervention-naïve major coronary segments (diameter ≥2.5 mm) determining a 40-70% diameter stenosis by visual assessment with no other significant stenosis (>70%) in the same vessel.
* Patient informed of the nature of the study, agreeing to it, and providing written informed consent as approved by the Ethics Committee of the respective clinical study site.
* Life expectancy >3 years.

Exclusion criteria:

* Female with childbearing potential or lactating.
* Acute or chronic renal dysfunction (defined as creatinine greater than 2.0 mg/dl).
* Advanced heart failure (NYHA III-IV)
* Stroke within the previous 6 months or spontaneous intracranial hemorrhage at any time.
* Severe valvular disease or valvular disease likely to require surgery or percutaneous valve replacement during the trial.
* Coronary anatomy preventing complete imaging of the segment of interest (including at least 5 mm at both stenosis edges).
* Lesions located in the left main coronary artery
* Diffusely diseased coronary artery segment or presence of ≥1 significant untreated non-culprit lesions (preventing correct adverse event attribution) in the coronary arteries.
* Prior myocardial infarction or coronary artery bypass graft [CABG] or PCI revascularization in the target coronary vessel.
* Coronary anatomy unsuitable for PCI.
* Comorbidities that might interfere with completion of the study procedures.
* Planned major surgery necessitating interruption of dual antiplatelet.
* Participating in another investigational drug or device trial that has not completed the primary endpoint or would interfere with the endpoints of this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1420 (Estimated)
Dates: Start 2021-06-30 (Actual); Primary Completion 2026-03-31 (Estimated); Study Completion 2028-03-31 (Estimated)

PRIMARY OUTCOMES:
Number of patients with cardiac death or non-fatal spontaneous target-vessel myocardial infarction | 2 years
  Composite outcome. Cardiac death will be defined as any death due to heart disease, including heart failure, myocardial infarction, arrhythmia, and sudden unexpected death.
  Any spontaneous myocardial infarction will be attributed to the randomized intermediate lesion if not clearly attributable to the non-target vessels.

SECONDARY OUTCOMES:
Number of patients with cardiac death | 2 years
  Cardiac death will be defined as any death due to heart disease, including heart failure, myocardial infarction, arrhythmia, and sudden unexpected death.
Number of patients with non-fatal spontaneous target-vessel Myocardial infarction (excluding peri-procedural MI) | 2 years
  Any spontaneous myocardial infarction will be attributed to the randomized intermediate lesion if not clearly attributable to the non-target vessels.
Number of patients with target lesion revascularization (either percutaneous or surgical) | 2 years
  Repeated lesion revascularization will be considered in case of repeated percutaneous coronary intervention and coronary artery bypass grafting the enrolled lesions.
Number of patients with composite of cardiac death and any myocardial infarction | 2 years
  Composite outcome. Cardiac death will be defined as any death due to heart disease, including heart failure, myocardial infarction, arrhythmia, and sudden unexpected death.
  Any spontaneous myocardial infarction will be collected regardless of the culprit vessel involved.
Number of patients with target vessel failure | 2 years
  Composite endpoint including cardiac death, non-fatal target-vessel MI, ischemia-driven target lesion revascularization.
Number of patients with composite endpoint of peri-procedural complications | Peri-procedural
  * contrast-induced nephropathy: a 25% increase in serum creatinine (SCr) from baseline or a 0.5 mg/dL (44 µmol/L) increase in absolute SCr value-within 48-72 hours after intravenous contrast administration.
  * dissection requiring bail-out stenting.
  * post-procedural MI: an increase within 48 hours after the index procedure of creatine kinase[CK]-MB (U/L) >5 times or Troponin (ng/L) >35 times above the normal value along with at least one of the followings: 1) symptoms of ischemia; 2) new or presumed new significant ST or T changes or new left bundle branch block; 3) new pathologic Q waves on an electrocardiogram; 4) new loss of viable myocardium or new regional wall motion abnormality; 5) reduced flow or major dissection in the coronary at angiography; or 6) intracoronary thrombus by angiography or autopsy.
  A stand-alone biomarker definition will be accepted in case of increase in the cardiac biomarker CK-MB >10 times or Troponin >70 times above the upper normal values.

CONTACTS AND LOCATIONS:
Overall Officials: Francesco Prati, MD, Principal Investigator — Centro per la Lotta con l'Infarto - CLI Foundation
Locations (34):
- University Hospital of Patras, Pátrai, AX, Greece
- Italy (29):
  - Ospedale C. e G. Mazzoni, Ascoli Piceno, AP
  - Ente ecclesiastico Ospedale Regionale Generale "F. Miulli", Acquaviva delle Fonti, BA
  - Policlinico University Hospital, Bari, BA
  - Di Venere Hospital, Bari, BA
  - ASST Papa Giovanni XXIII, Bergamo, BG
  - Azienda Ospedaliera San Pio, Benevento, BN
  - Azienda Ospedaliero_Universitaria IRCCS Policlinico di St.Orsola, Bologna, BO
  - ARNAS Brotzu, Cagliari, CA
  - P.O. San Giuseppe Moscati, Aversa, CE
  - Azienda Ospedaliera "Policlinico "G. Rodolico- San Marco", Catania, CT
  - Azienda Ospedaliera Per L'emergenza Cannizzaro, Catania, CT
  - IRCCS Casa sollievo della sofferenza, San Giovanni Rotondo, FG
  - IRCCS Ospedale Policlinico San Martino, Genova, GE
  - Misericordia Hospital, Grosseto, GR
  - Ospedale Vito Fazzi, Lecce, LE
  - Ospedale Santa Maria Goretti, Latina, Latina, LT
  - Azienda Ospedaliero Universitaria Policlinico "G. Martino", Messina, Messina, ME
  - Centro Cardiologico Monzino IRCCS, Milan, MI
  - IRCCS Galeazzi- Sant'Ambrogio, Milan, MI
  - San Camillo Hospital, Roma, RM
  - Fondazione Policlinico Universitario Agostino Gemelli IRCCS, Roma, RM
  - UOSA Cardiologia Interventistica, Siena, SI
  - P.O. Umberto I, Syracuse, SR
  - Struttura Complessa di Cardiologia Clinica e Interventistica, Sassari, SS
  - Rivoli Hospital, Rivoli, TO
  - Ospedale Conegliano, Conegliano, TV
  - Azienda Sanitaria Universitaria Friuli Centrale - Udine University Hospital, Udine, UD
  - Federico II di Napoli, Napoli
  - San Giovanni Hospital, Rome
- Spain (3):
  - Hospital Virgen de la Victoria, Málaga, MA
  - Hospital universitario La Princesa, Madrid, Madrid, M
  - Hospital Universitario Central de Asturias, Oviedo
- Inselspital, Bern University Hospital, Bern, Canton of Bern, Switzerland

IPD SHARING:
Plan to Share IPD: Yes
After the publication of the main paper, anonymized data will be shared upon reasonable request after discussion by the Steering Committee.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: After the publication of the main paper
Access Criteria: Anonymised data will be shared upon reasonable request, after discussion by the Steering Committee.

REFERENCES:
- [Background] Tonino PA, Fearon WF, De Bruyne B, Oldroyd KG, Leesar MA, Ver Lee PN, Maccarthy PA, Van't Veer M, Pijls NH. Angiographic versus functional severity of coronary artery stenoses in the FAME study fractional flow reserve versus angiography in multivessel evaluation. J Am Coll Cardiol. 2010 Jun 22;55(25):2816-21. doi: 10.1016/j.jacc.2009.11.096. PMID 20579537
- [Background] Toth G, Hamilos M, Pyxaras S, Mangiacapra F, Nelis O, De Vroey F, Di Serafino L, Muller O, Van Mieghem C, Wyffels E, Heyndrickx GR, Bartunek J, Vanderheyden M, Barbato E, Wijns W, De Bruyne B. Evolving concepts of angiogram: fractional flow reserve discordances in 4000 coronary stenoses. Eur Heart J. 2014 Oct 21;35(40):2831-8. doi: 10.1093/eurheartj/ehu094. Epub 2014 Mar 18. PMID 24644308
- [Background] Pijls NH, van Schaardenburgh P, Manoharan G, Boersma E, Bech JW, van't Veer M, Bar F, Hoorntje J, Koolen J, Wijns W, de Bruyne B. Percutaneous coronary intervention of functionally nonsignificant stenosis: 5-year follow-up of the DEFER Study. J Am Coll Cardiol. 2007 May 29;49(21):2105-11. doi: 10.1016/j.jacc.2007.01.087. Epub 2007 May 17. PMID 17531660
- [Background] Tonino PA, De Bruyne B, Pijls NH, Siebert U, Ikeno F, van' t Veer M, Klauss V, Manoharan G, Engstrom T, Oldroyd KG, Ver Lee PN, MacCarthy PA, Fearon WF; FAME Study Investigators. Fractional flow reserve versus angiography for guiding percutaneous coronary intervention. N Engl J Med. 2009 Jan 15;360(3):213-24. doi: 10.1056/NEJMoa0807611. PMID 19144937
- [Background] Burzotta F, Leone AM, Aurigemma C, Zambrano A, Zimbardo G, Arioti M, Vergallo R, De Maria GL, Cerracchio E, Romagnoli E, Trani C, Crea F. Fractional Flow Reserve or Optical Coherence Tomography to Guide Management of Angiographically Intermediate Coronary Stenosis: A Single-Center Trial. JACC Cardiovasc Interv. 2020 Jan 13;13(1):49-58. doi: 10.1016/j.jcin.2019.09.034. PMID 31918942
- [Background] Waksman R, Legutko J, Singh J, Orlando Q, Marso S, Schloss T, Tugaoen J, DeVries J, Palmer N, Haude M, Swymelar S, Torguson R. FIRST: Fractional Flow Reserve and Intravascular Ultrasound Relationship Study. J Am Coll Cardiol. 2013 Mar 5;61(9):917-23. doi: 10.1016/j.jacc.2012.12.012. Epub 2013 Jan 23. PMID 23352786
- [Background] Cho YK, Nam CW, Han JK, Koo BK, Doh JH, Ben-Dor I, Waksman R, Pichard A, Murata N, Tanaka N, Lee CH, Gonzalo N, Escaned J, Costa MA, Kubo T, Akasaka T, Hu X, Wang JA, Yang HM, Yoon MH, Tahk SJ, Yoon HJ, Chung IS, Hur SH, Kim KB. Usefulness of combined intravascular ultrasound parameters to predict functional significance of coronary artery stenosis and determinants of mismatch. EuroIntervention. 2015 Jun;11(2):163-70. doi: 10.4244/EIJV11I2A30. PMID 26093837
- [Background] Usui E, Yonetsu T, Kanaji Y, Hoshino M, Yamaguchi M, Hada M, Hamaya R, Kanno Y, Murai T, Lee T, Kakuta T. Efficacy of Optical Coherence Tomography-derived Morphometric Assessment in Predicting the Physiological Significance of Coronary Stenosis: Head-to-Head Comparison with Intravascular Ultrasound. EuroIntervention. 2018 Apr 6;13(18):e2210-e2218. doi: 10.4244/EIJ-D-17-00613. PMID 29155383
- [Background] D'Ascenzo F, Barbero U, Cerrato E, Lipinski MJ, Omede P, Montefusco A, Taha S, Naganuma T, Reith S, Voros S, Latib A, Gonzalo N, Quadri G, Colombo A, Biondi-Zoccai G, Escaned J, Moretti C, Gaita F. Accuracy of intravascular ultrasound and optical coherence tomography in identifying functionally significant coronary stenosis according to vessel diameter: A meta-analysis of 2,581 patients and 2,807 lesions. Am Heart J. 2015 May;169(5):663-73. doi: 10.1016/j.ahj.2015.01.013. Epub 2015 Feb 21. PMID 25965714
- [Background] Prati F, Romagnoli E, Gatto L, La Manna A, Burzotta F, Ozaki Y, Marco V, Boi A, Fineschi M, Fabbiocchi F, Taglieri N, Niccoli G, Trani C, Versaci F, Calligaris G, Ruscica G, Di Giorgio A, Vergallo R, Albertucci M, Biondi-Zoccai G, Tamburino C, Crea F, Alfonso F, Arbustini E. Relationship between coronary plaque morphology of the left anterior descending artery and 12 months clinical outcome: the CLIMA study. Eur Heart J. 2020 Jan 14;41(3):383-391. doi: 10.1093/eurheartj/ehz520. PMID 31504405
- [Background] Stone GW, Maehara A, Lansky AJ, de Bruyne B, Cristea E, Mintz GS, Mehran R, McPherson J, Farhat N, Marso SP, Parise H, Templin B, White R, Zhang Z, Serruys PW; PROSPECT Investigators. A prospective natural-history study of coronary atherosclerosis. N Engl J Med. 2011 Jan 20;364(3):226-35. doi: 10.1056/NEJMoa1002358. PMID 21247313
- [Background] Di Vito L, Agozzino M, Marco V, Ricciardi A, Concardi M, Romagnoli E, Gatto L, Calogero G, Tavazzi L, Arbustini E, Prati F. Identification and quantification of macrophage presence in coronary atherosclerotic plaques by optical coherence tomography. Eur Heart J Cardiovasc Imaging. 2015 Jul;16(7):807-13. doi: 10.1093/ehjci/jeu307. Epub 2015 Jan 14. PMID 25588802

DOCUMENTS (1):
  • Informed Consent Form (2025-02-15): https://cdn.clinicaltrials.gov/large-docs/84/NCT05027984/ICF_001.pdf